CLINICAL TRIAL: NCT03824691
Title: Cabozantinib Plus Durvalumab in Patients With Advanced and Chemotherapy-treated Bladder Carcinoma, of Urothelial and Non-urothelial Histology: an Open-label, Single-centre, Phase 2, Single-arm Proof-of-concept Trial: ARCADIA Study
Brief Title: hARnessing CAbozantinib and Durvalumab Immuno-oncology Association: ARCADIA Study"
Acronym: ARCADIA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INT 180/18
Record Dates: First submitted 2019-01-08; First posted 2019-01-31 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Bladder Carcinoma
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — cabozantinib; durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cabozantinib + Durvalumab (Experimental): Subjects will receive 1500 mg durvalumab (MEDI4736) IV infusion every 28 days + Cabozantinib 40 mg orally once daily
  Interventions: Drug: Cabozantinib; Drug: Durvalumab

INTERVENTIONS:
Drug: Cabozantinib — cabozantinib 40 mg orally once daily
  Other Names: CABOMETYX
Drug: Durvalumab — 1500 mg durvalumab (MEDI4736) IV infusion every 28 days
  Other Names: Imfinzi

SUMMARY:
Cabozantinib plus Durvalumab in patients with advanced and chemotherapy-treated bladder carcinoma, of urothelial and non-urothelial histology: an open-label, single-centre, phase 2, single-arm proof-of-concept trial: ARCADIA study

DETAILED DESCRIPTION:
an open-label, single-centre, phase 2,

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent.
* Age ≥18 years.
* Body weight >30kg
* Histologically-confirmed diagnosis of UC or variant histologies (e.g. squamous cell carcinoma, adenocarcinoma, micropapillary tumors, BUT excluding pure small cell carcinoma) of the bladder or the urothelium.
* Either bladder, urethral, or upper tract primary tumor will be allowed.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
* Life expectancy of at ≥ 12 weeks.
* Availability of tumor tissue for PD-L1 IHC assay.
* Measurable and non-measurable disease will be included (e.g. patients with bone metastases only will be allowed for inclusion).
* Failure of 1 or 2 cisplatin-based conventional chemotherapy regimens for metastatic disease (2nd-to-3rd line only).
* Neoadjuvant/adjuvant regimens will be counted provided that a relapse occurred with 6 months of the last cycle of chemotherapy.
* Adequate function of the organs:

  1. Absolute neutrophil count (ANC) ≥ 1500/mm3
  2. Platelets ≥ 100,000/mm3
  3. Hemoglobin ≥ 9 g/dL (≥ 90 g/L).
  4. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 3.0 × upper limit of normal.
  5. Total bilirubin ≤ 1.5 × the upper limit of normal. For subjects with Gilbert's disease ≤ 3 mg/dL

  g. Serum creatinine ≤ 2.0 × upper limit of normal or calculated creatinine clearance ≥ 30 mL/min using the Cockroft-Gault equation h. Lipase < 2.0 times the upper limit of normal (ULN)
* Recovery to baseline or ≤ Grade 1 Common Terminology Criteria for Adverse Events (CTCAE) v5.0 from toxicities related to any prior treatments, unless AE(s) are clinically nonsignificant and/or stable on supportive therapy
* Ability to swallow tablets
* Contraception for sexually active fertile patients and their partners. Of note, a barrier method is recommended in addition to the use of steroid hormonal contraceptives, because the effects of cabozantinib on the pharmacokinetics of the latter are unknown.
* Evidence of post menopausal status or serum pregnancy test for female pre-menopausal subject

Exclusion Criteria:

* Patients taking regular oral steroids, above the allowed limit of 10mg/day methylprednisolone or analogues, for any reason. Patients must not have had steroids for 28 days prior to study entry.
* Malignancies other than bladder carcinoma within 5 years prior to Cycle 1, Day 1, with the exception of those with a negligible risk of metastasis or death and treated with expected curative outcome (such as adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer, or ductal carcinoma in situ treated surgically with curative intent) or localized prostate cancer treated with curative intent and absence of prostate-specific antigen (PSA) relapse or incidental prostate cancer (Gleason score ≤ 3 + 4 and PSA < 10 ng/mL undergoing active surveillance and treatment naive).
* Evidence of significant uncontrolled concomitant disease that could affect compliance with the protocol or interpretation of results.
* Active or untreated CNS metastases as determined by computed tomography (CT) or magnetic resonance imaging evaluation during screening and prior radiographic assessments.
* Patients with treated asymptomatic CNS metastases are eligible, provided they meet all of the following criteria:

  1. Evaluable or measurable disease outside the CNS
  2. No metastases to midbrain, pons, medulla, or within 10 mm of the optic apparatus (optic nerves and chiasm)
  3. No history of intracranial or spinal cord hemorrhage
  4. No ongoing requirement for corticosteroid as therapy for CNS disease; anti-convulsants at a stable dose are allowed
  5. No evidence of significant vasogenic edema
  6. No stereotactic radiation, whole-brain radiation or neurosurgical resection within 4 weeks prior to Cycle 1, Day 1
  7. Radiographic demonstration of interim stability (i.e., no progression) between the completion of CNS-directed therapy and the screening radiographic study
  8. Screening CNS radiographic study ≥ 4 weeks since completion of radiotherapy or surgical resection and ≥ 2 weeks since discontinuation of corticosteroids
* Pregnant female patients. All female patients of childbearing potential with a positive pregnancy test within 2 weeks prior to the first dose of study treatment will be excluded from the study.
* Clinically significant cardiovascular disease, for example, myocardial infarction (within 3months prior to enrolment), unstable angina, New York Heart Association (NYHA) grade II or greater congestive heart failure or serious cardiac arrhythmia requiring medication (beta-blockers and digoxin are allowed)
* Uncontrolled hypertension, stroke or other ischemic or thromboembolic event (DVT, PE) within 6 months before first dose of cabozantinib.
* Severe infections within 4 weeks prior to enrolment in the study including but not limited to hospitalization for complications of infection, bacteraemia, or severe pneumonia.
* Major surgical procedure within 4 weeks prior to enrolmentor anticipation of need for a major surgical procedure during the course of the study other than for diagnosis. Complete wound healing from major surgery must have occurred 1 month before inclusion and from minor surgery (eg, simple excision, tooth extraction) at least 10 days before inclusion. Subjects with clinically relevant ongoing complications from prior surgery are not eligible.
* Received therapeutic oral or intravenous (IV) antibiotics within 2 weeks prior to enrolment (patients receiving prophylactic antibiotics, e.g., for prevention of a urinary tract infection or chronic obstructive pulmonary disease, are eligible).
* Concomitant anticoagulation with oral anticoagulants or platelet inhibitors.
* History of autoimmune disease including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis.
* Patients with a history of autoimmune-related hypothyroidism, unless on a stable dose of thyroid-replacement hormone.
* Patients with uncontrolled Type 1 diabetes mellitus
* Uncontrolled hypercalcemia (> 1.5 mmol/L ionized calcium or Ca > 12 mg/dL or corrected serum calcium > ULN) or symptomatic hypercalcemia requiring continued use of bisphosphonate therapy or denosumab. Patients who are receiving bisphosphonate therapy or denosumab specifically to prevent skeletal events and who do not have a history of clinically significant hypercalcemia are eligible. Patients who are receiving denosumab prior to enrollment must be willing and eligible to receive a bisphosphonate instead while on study.
* radiation therapy for bone within 2 weeks or other radiation therapy within 4 weeks before first dose of study treatment. patients with clinically relevant ongoing complications from prior radiation therapy
* serious non healing wound/ulcer/bone fracture, moderate to severe hepatic impairment (Child Pugh B or C)
* History of idiopathic pulmonary fibrosis (including pneumonitis), drug-induced pneumonitis, organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia), or evidence of active pneumonitis on screening chest CT scan (History of radiation pneumonitis in the radiation field (fibrosis) is permitted).
* Patients with tumors invading major pulmonary vessels and/or with cavitating pulmonary lesions.
* Positive test for HIV.
* Patients with active hepatitis infection (defined as having a positive hepatitis B surface antigen [HBsAg] test at screening) or hepatitis C. Patients with past hepatitis B virus (HBV) infection or resolved HBV infection (defined as having a negative HBs Ag test and a positive antibody to hepatitis B core antigen [anti-HBc] antibody test) are eligible. Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV RNA.
* Patients with active tuberculosis.
* Gastrointestinal disorders likely to interfere with absorption of the study drug (e.g. partial bowel obstruction or malabsorption).
* Subjects with gastrointestinal disorders associated with a high risk of perforation or fistula formation
* Subjects with active peptic ulcer or with a history of clinically significant GI bleeding within 12 weeks before the first dose of study treatment
* Prior treatment with CD137 agonists, anti-PD-1, or anti-PD-L1 therapeutic antibody or pathway-targeting agents.
* Administration of a live, attenuated vaccine within 4 weeks prior to enrolment or anticipation that such a live, attenuated vaccine will be required during the study.
* Treatment with any other investigational agent or participation in another clinical trial with therapeutic intent within 28 days prior to enrolment.
* Treatment with systemic immunostimulatory agents (including but not limited to interferons or interleukin [IL]-2) within 4 weeks or five half-lives of the drug, whichever is shorter, prior to enrolment.
* Rare hereditary problems of galactose intolerance, the Lapp lactase deficiency or glucose-galactose malabsorption

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2019-09-25 (Actual); Primary Completion 2023-02 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint of the study will be overall survival (OS). | 48 months
  to evaluate whether the combination of durvalumab and cabozantinib will be active and will result in an increased efficacy compared to the available results with the use of both single-agents

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability). | 48 months
  incidence, nature and severity of all-cause and treatment-related adverse events (AE), graded with the Common Terminology Criteria for Adverse Events (CTCAE), version 5.0.
progression-free survival (PFS) | 48 months
  RECIST 1.1 criteria
responses to treatment | 48 months
  Assessment of RR (investigator-assessed) according to the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria. RR (%) = complete (CR) + partial responses (PR)
response duration | 48 months
  PET-responses according to the EORTC criteria
Biomarkers of activity and efficacy of either agents and their combination. | 48 months
  determination of a patient's PD-L1 status. Biomarkers Blood Collection will be performend at baseline, every 2 cycles and progression disease

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Istituto Nazionale Tumori, Milan, Italy

REFERENCES:
- [Result] Kamat AM, Hahn NM, Efstathiou JA, Lerner SP, Malmstrom PU, Choi W, Guo CC, Lotan Y, Kassouf W. Bladder cancer. Lancet. 2016 Dec 3;388(10061):2796-2810. doi: 10.1016/S0140-6736(16)30512-8. Epub 2016 Jun 23. PMID 27345655
- [Result] Necchi A, Sonpavde G, Lo Vullo S, Giardiello D, Bamias A, Crabb SJ, Harshman LC, Bellmunt J, De Giorgi U, Sternberg CN, Cerbone L, Ladoire S, Wong YN, Yu EY, Chowdhury S, Niegisch G, Srinivas S, Vaishampayan UN, Pal SK, Agarwal N, Alva A, Baniel J, Golshayan AR, Morales-Barrera R, Bowles DW, Milowsky MI, Theodore C, Berthold DR, Daugaard G, Sridhar SS, Powles T, Rosenberg JE, Galsky MD, Mariani L; RISC Investigators. Nomogram-based Prediction of Overall Survival in Patients with Metastatic Urothelial Carcinoma Receiving First-line Platinum-based Chemotherapy: Retrospective International Study of Invasive/Advanced Cancer of the Urothelium (RISC). Eur Urol. 2017 Feb;71(2):281-289. doi: 10.1016/j.eururo.2016.09.042. Epub 2016 Oct 8. PMID 27726966
- [Result] Raggi D, Miceli R, Sonpavde G, Giannatempo P, Mariani L, Galsky MD, Bellmunt J, Necchi A. Second-line single-agent versus doublet chemotherapy as salvage therapy for metastatic urothelial cancer: a systematic review and meta-analysis. Ann Oncol. 2016 Jan;27(1):49-61. doi: 10.1093/annonc/mdv509. Epub 2015 Oct 20. PMID 26487582
- [Result] Necchi A, Pond GR, Raggi D, Giannatempo P, Vogelzang NJ, Grivas P, Galsky MD, Bellmunt J, Sonpavde G. Efficacy and Safety of Gemcitabine Plus Either Taxane or Carboplatin in the First-Line Setting of Metastatic Urothelial Carcinoma: A Systematic Review and Meta-Analysis. Clin Genitourin Cancer. 2017 Feb;15(1):23-30.e2. doi: 10.1016/j.clgc.2016.05.003. Epub 2016 May 27. PMID 27324051
- [Result] Dash A, Galsky MD, Vickers AJ, Serio AM, Koppie TM, Dalbagni G, Bochner BH. Impact of renal impairment on eligibility for adjuvant cisplatin-based chemotherapy in patients with urothelial carcinoma of the bladder. Cancer. 2006 Aug 1;107(3):506-13. doi: 10.1002/cncr.22031. PMID 16773629
- [Result] Galsky MD, Hahn NM, Rosenberg J, Sonpavde G, Hutson T, Oh WK, Dreicer R, Vogelzang N, Sternberg CN, Bajorin DF, Bellmunt J. Treatment of patients with metastatic urothelial cancer "unfit" for Cisplatin-based chemotherapy. J Clin Oncol. 2011 Jun 10;29(17):2432-8. doi: 10.1200/JCO.2011.34.8433. Epub 2011 May 9. PMID 21555688
- [Result] Reardon ZD, Patel SG, Zaid HB, Stimson CJ, Resnick MJ, Keegan KA, Barocas DA, Chang SS, Cookson MS. Trends in the use of perioperative chemotherapy for localized and locally advanced muscle-invasive bladder cancer: a sign of changing tides. Eur Urol. 2015 Jan;67(1):165-170. doi: 10.1016/j.eururo.2014.01.009. Epub 2014 Jan 23. PMID 24472710
- [Result] Gentzler R, Hall R, Kunk PR, Gaughan E, Dillon P, Slingluff CL Jr, Rahma OE. Beyond melanoma: inhibiting the PD-1/PD-L1 pathway in solid tumors. Immunotherapy. 2016 May;8(5):583-600. doi: 10.2217/imt-2015-0029. PMID 27140411
- [Result] Powles T, Eder JP, Fine GD, Braiteh FS, Loriot Y, Cruz C, Bellmunt J, Burris HA, Petrylak DP, Teng SL, Shen X, Boyd Z, Hegde PS, Chen DS, Vogelzang NJ. MPDL3280A (anti-PD-L1) treatment leads to clinical activity in metastatic bladder cancer. Nature. 2014 Nov 27;515(7528):558-62. doi: 10.1038/nature13904. PMID 25428503
- [Result] Herr HW, Morales A. History of bacillus Calmette-Guerin and bladder cancer: an immunotherapy success story. J Urol. 2008 Jan;179(1):53-6. doi: 10.1016/j.juro.2007.08.122. Epub 2007 Nov 13. PMID 17997439
- [Result] Rink M, Shariat SF, Soave A. Liquid biopsies in bladder cancer-did we find the Holy Grail for biomarker analyses? Transl Androl Urol. 2016 Dec;5(6):980-983. doi: 10.21037/tau.2016.09.03. No abstract available. PMID 28078238
- [Result] Cancer Genome Atlas Research Network. Comprehensive molecular characterization of urothelial bladder carcinoma. Nature. 2014 Mar 20;507(7492):315-22. doi: 10.1038/nature12965. Epub 2014 Jan 29. PMID 24476821
- [Result] Lawrence MS, Stojanov P, Polak P, Kryukov GV, Cibulskis K, Sivachenko A, Carter SL, Stewart C, Mermel CH, Roberts SA, Kiezun A, Hammerman PS, McKenna A, Drier Y, Zou L, Ramos AH, Pugh TJ, Stransky N, Helman E, Kim J, Sougnez C, Ambrogio L, Nickerson E, Shefler E, Cortes ML, Auclair D, Saksena G, Voet D, Noble M, DiCara D, Lin P, Lichtenstein L, Heiman DI, Fennell T, Imielinski M, Hernandez B, Hodis E, Baca S, Dulak AM, Lohr J, Landau DA, Wu CJ, Melendez-Zajgla J, Hidalgo-Miranda A, Koren A, McCarroll SA, Mora J, Crompton B, Onofrio R, Parkin M, Winckler W, Ardlie K, Gabriel SB, Roberts CWM, Biegel JA, Stegmaier K, Bass AJ, Garraway LA, Meyerson M, Golub TR, Gordenin DA, Sunyaev S, Lander ES, Getz G. Mutational heterogeneity in cancer and the search for new cancer-associated genes. Nature. 2013 Jul 11;499(7457):214-218. doi: 10.1038/nature12213. Epub 2013 Jun 16. PMID 23770567
- [Result] Massard C, Gordon MS, Sharma S, Rafii S, Wainberg ZA, Luke J, Curiel TJ, Colon-Otero G, Hamid O, Sanborn RE, O'Donnell PH, Drakaki A, Tan W, Kurland JF, Rebelatto MC, Jin X, Blake-Haskins JA, Gupta A, Segal NH. Safety and Efficacy of Durvalumab (MEDI4736), an Anti-Programmed Cell Death Ligand-1 Immune Checkpoint Inhibitor, in Patients With Advanced Urothelial Bladder Cancer. J Clin Oncol. 2016 Sep 10;34(26):3119-25. doi: 10.1200/JCO.2016.67.9761. Epub 2016 Jun 6. PMID 27269937
- [Result] Powles T, O'Donnell PH, Massard C, Arkenau HT, Friedlander TW, Hoimes CJ, Lee JL, Ong M, Sridhar SS, Vogelzang NJ, Fishman MN, Zhang J, Srinivas S, Parikh J, Antal J, Jin X, Gupta AK, Ben Y, Hahn NM. Efficacy and Safety of Durvalumab in Locally Advanced or Metastatic Urothelial Carcinoma: Updated Results From a Phase 1/2 Open-label Study. JAMA Oncol. 2017 Sep 14;3(9):e172411. doi: 10.1001/jamaoncol.2017.2411. Epub 2017 Sep 14. PMID 28817753
- [Result] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774
- [Result] Seymour L, Bogaerts J, Perrone A, Ford R, Schwartz LH, Mandrekar S, Lin NU, Litiere S, Dancey J, Chen A, Hodi FS, Therasse P, Hoekstra OS, Shankar LK, Wolchok JD, Ballinger M, Caramella C, de Vries EGE; RECIST working group. iRECIST: guidelines for response criteria for use in trials testing immunotherapeutics. Lancet Oncol. 2017 Mar;18(3):e143-e152. doi: 10.1016/S1470-2045(17)30074-8. Epub 2017 Mar 2. PMID 28271869
- [Result] Young H, Baum R, Cremerius U, Herholz K, Hoekstra O, Lammertsma AA, Pruim J, Price P. Measurement of clinical and subclinical tumour response using [18F]-fluorodeoxyglucose and positron emission tomography: review and 1999 EORTC recommendations. European Organization for Research and Treatment of Cancer (EORTC) PET Study Group. Eur J Cancer. 1999 Dec;35(13):1773-82. doi: 10.1016/s0959-8049(99)00229-4. PMID 10673991
- [Result] Zehir A, Benayed R, Shah RH, Syed A, Middha S, Kim HR, Srinivasan P, Gao J, Chakravarty D, Devlin SM, Hellmann MD, Barron DA, Schram AM, Hameed M, Dogan S, Ross DS, Hechtman JF, DeLair DF, Yao J, Mandelker DL, Cheng DT, Chandramohan R, Mohanty AS, Ptashkin RN, Jayakumaran G, Prasad M, Syed MH, Rema AB, Liu ZY, Nafa K, Borsu L, Sadowska J, Casanova J, Bacares R, Kiecka IJ, Razumova A, Son JB, Stewart L, Baldi T, Mullaney KA, Al-Ahmadie H, Vakiani E, Abeshouse AA, Penson AV, Jonsson P, Camacho N, Chang MT, Won HH, Gross BE, Kundra R, Heins ZJ, Chen HW, Phillips S, Zhang H, Wang J, Ochoa A, Wills J, Eubank M, Thomas SB, Gardos SM, Reales DN, Galle J, Durany R, Cambria R, Abida W, Cercek A, Feldman DR, Gounder MM, Hakimi AA, Harding JJ, Iyer G, Janjigian YY, Jordan EJ, Kelly CM, Lowery MA, Morris LGT, Omuro AM, Raj N, Razavi P, Shoushtari AN, Shukla N, Soumerai TE, Varghese AM, Yaeger R, Coleman J, Bochner B, Riely GJ, Saltz LB, Scher HI, Sabbatini PJ, Robson ME, Klimstra DS, Taylor BS, Baselga J, Schultz N, Hyman DM, Arcila ME, Solit DB, Ladanyi M, Berger MF. Mutational landscape of metastatic cancer revealed from prospective clinical sequencing of 10,000 patients. Nat Med. 2017 Jun;23(6):703-713. doi: 10.1038/nm.4333. Epub 2017 May 8. PMID 28481359
- [Derived] Marandino L, Raggi D, Calareso G, Alessi A, Colecchia M, Martini A, Briganti A, Montorsi F, Madison R, Ross JS, Necchi A. Cabozantinib Plus Durvalumab in Patients With Advanced Urothelial Carcinoma After Platinum Chemotherapy: Safety and Preliminary Activity of the Open-Label, Single-Arm, Phase 2 ARCADIA Trial. Clin Genitourin Cancer. 2021 Oct;19(5):457-465. doi: 10.1016/j.clgc.2021.04.001. Epub 2021 Apr 21. PMID 34006499